CLINICAL TRIAL: NCT01524133
Title: Randomized Trial of Sertraline, Prolonged Exposure, and Their Combination for Post-traumatic Stress Disorder (PTSD) in Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF).
Brief Title: PROlonGed ExpoSure Sertraline
Acronym: PROGrESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sheila Rauch, Clinical Director of Wounded Warrior Project and Associate Professor at Emory University, Principal Investigator, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROGrESS
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: combat-related PTSD; Posttraumatic stress disorder; prolonged exposure therapy; sertraline; military; veterans; VA hospital; mental illness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Mental Disorders | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sertraline + enhanced medication management (SERT/EMM) (Active Comparator): 24 weeks of sertraline + enhanced medication management
  Interventions: Drug: Sertraline
- Prolonged Exposure + sertraline (PE/SERT) (Active Comparator): Up to 13 sessions of prolonged exposure therapy + 24 weeks of sertraline
  Interventions: Drug: Sertraline; Behavioral: Prolonged Exposure Therapy
- Prolonged Exposure + placebo (PE/PLB) (Active Comparator): Up to 13 sessions of prolonged exposure therapy + 24 weeks of placebo
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Drug: Sertraline — Initial baseline dose of 25 mg/day. Clinician will attempt to titrate patients to at least 100 mg/day and up to 200 mg/day if tolerated by week 8.
  Other Names: Zoloft
  Arms: Prolonged Exposure + sertraline (PE/SERT); Sertraline + enhanced medication management (SERT/EMM)
Behavioral: Prolonged Exposure Therapy — up to 13 sessions of prolonged exposure
  Arms: Prolonged Exposure + placebo (PE/PLB); Prolonged Exposure + sertraline (PE/SERT)

SUMMARY:
The current research study aims to compare the effectiveness of two proven treatments for posttraumatic stress disorder (PTSD): Prolonged Exposure (PE), sertraline, and their combination. In addition, the investigators are examining predictors of response to these two treatments and how PTSD symptoms, thoughts, and biological factors may be changed by such treatments. Biological mechanisms of change are also examined including emotion processing and regulation in fMRI, HPA axis function, and genetics and genomics. In addition, the investigators will examine acceptability of each treatment and reasons for ending treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn (OEF/OIF/OND) combat veteran with chronic posttraumatic stress disorder (PTSD) or significant PTSD symptoms (Clinician Administered Posttraumatic Stress Disorder Scale [CAPS] >= 50) of at least 3 months duration

Exclusion Criteria:

* Current, imminent risk of suicide (as indicated on C-SSRS)
* Active psychosis
* Alcohol or substance dependence in the past 8 weeks
* Unable to attend regular appointments
* Prior intolerance or failure of adequate trial of prolonged exposure (PE) or sertraline (SERT) (defined as at least 2 months of SERT at least 100mg/day)
* Medical illness likely to result in hospitalization or for which treatments are contraindicated (based on lab results, medical history and physical exam)
* Serious cognitive impairment (as evidenced by cognitive impairment felt likely to interfere with the ability to participate meaningfully in the study)
* Concurrent antidepressants or antipsychotics
* Pregnant females

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2011-11; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Rauch, PhD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (4):
- United States (4):
  - VA San Diego Healthcare System, San Diego, California
  - Ralph H. Johnson VA Medical Center/Savannah Primary Care Clinic, Savannah, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Veterans Affairs Ann Arbor Healthcare System, Ann Arbor, Michigan

REFERENCES:
- [Derived] Allard CB, Norman SB, Straus E, Kim HM, Stein MB, Simon NM, Rauch SAM; PROGrESS Study Team. Reductions in guilt cognitions following prolonged exposure and/or sertraline predict subsequent improvements in PTSD and depression. J Behav Ther Exp Psychiatry. 2021 Dec;73:101666. doi: 10.1016/j.jbtep.2021.101666. Epub 2021 Jun 1. PMID 34147766
- [Derived] Rauch SAM, Kim HM, Lederman S, Sullivan G, Acierno R, Tuerk PW, Simon NM, Venners MR, Norman SB, Allard CB, Porter KE, Martis B, Bui E, Baker AW; PROGrESS Team. Predictors of Response to Prolonged Exposure, Sertraline, and Their Combination for the Treatment of Military PTSD. J Clin Psychiatry. 2021 Jun 15;82(4):20m13752. doi: 10.4088/JCP.20m13752. PMID 34133087
- [Derived] Sheynin J, Duval ER, King AP, Angstadt M, Phan KL, Simon NM, Rauch SAM, Liberzon I. Associations between resting-state functional connectivity and treatment response in a randomized clinical trial for posttraumatic stress disorder. Depress Anxiety. 2020 Oct;37(10):1037-1046. doi: 10.1002/da.23075. Epub 2020 Jul 15. PMID 32668087
- [Derived] Rauch SAM, King A, Kim HM, Powell C, Rajaram N, Venners M, Simon NM, Hamner M, Liberzon I. Cortisol awakening response in PTSD treatment: Predictor or mechanism of change. Psychoneuroendocrinology. 2020 Aug;118:104714. doi: 10.1016/j.psyneuen.2020.104714. Epub 2020 May 15. PMID 32446108
- [Derived] Duval ER, Sheynin J, King AP, Phan KL, Simon NM, Martis B, Porter KE, Norman SB, Liberzon I, Rauch SAM. Neural function during emotion processing and modulation associated with treatment response in a randomized clinical trial for posttraumatic stress disorder. Depress Anxiety. 2020 Jul;37(7):670-681. doi: 10.1002/da.23022. Epub 2020 Apr 19. PMID 32306485
- [Derived] Joshi SA, Duval ER, Sheynin J, King AP, Phan KL, Martis B, Porter KE, Liberzon I, Rauch SAM. Neural correlates of emotional reactivity and regulation associated with treatment response in a randomized clinical trial for posttraumatic stress disorder. Psychiatry Res Neuroimaging. 2020 May 30;299:111062. doi: 10.1016/j.pscychresns.2020.111062. Epub 2020 Mar 5. PMID 32278278
- [Derived] Goetter EM, Hoeppner SS, Khan AJ, Charney ME, Wieman S, Venners MR, Avallone KM, Rauch SAM, Simon NM. Combat-Related Posttraumatic Stress Disorder and Comorbid Major Depression in U.S. Veterans: The Role of Deployment Cycle Adversity and Social Support. J Trauma Stress. 2020 Jun;33(3):276-284. doi: 10.1002/jts.22496. Epub 2020 Mar 26. PMID 32216142
- [Derived] Rauch SAM, Kim HM, Powell C, Tuerk PW, Simon NM, Acierno R, Allard CB, Norman SB, Venners MR, Rothbaum BO, Stein MB, Porter K, Martis B, King AP, Liberzon I, Phan KL, Hoge CW. Efficacy of Prolonged Exposure Therapy, Sertraline Hydrochloride, and Their Combination Among Combat Veterans With Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Feb 1;76(2):117-126. doi: 10.1001/jamapsychiatry.2018.3412. PMID 30516797
- [Derived] Rauch SAM, Simon NM, Kim HM, Acierno R, King AP, Norman SB, Venners MR, Porter K, Phan KL, Tuerk PW, Allard C, Liberzon I, Rothbaum BO, Martis B, Stein MB, Hoge CW. Integrating biological treatment mechanisms into randomized clinical trials: Design of PROGrESS (PROlonGed ExpoSure and Sertraline Trial). Contemp Clin Trials. 2018 Jan;64:128-138. doi: 10.1016/j.cct.2017.10.013. Epub 2017 Oct 29. PMID 29081351

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were informed of assignment at first treatment visit. Only those randomized patients who started treatment are included below (16 patients never started treatment. They did not know condition assignment.).
Period: Treatment Phase
Arm/Group | Sertraline + Enhanced Medication Management (SERT/EMM) | Prolonged Exposure + Sertraline (PE/SERT) | Prolonged Exposure + Placebo (PE/PLB)
Started | 71 | 69 | 67
Completed | 52 (Completed Both Assigned treatment) | 37 (Completed Both Assigned Treatments) | 31 (Completed both assigned treatments)
Not Completed | 19 | 32 | 36
Not completed — Withdrawal by Subject | 13 | 28 | 31
Not completed — Physician Decision | 6 | 3 | 3
Not completed — Lost to Follow-up | 0 | 1 | 2
Period: Overall Study 52 Weeks
Arm/Group | Sertraline + Enhanced Medication Management (SERT/EMM) | Prolonged Exposure + Sertraline (PE/SERT) | Prolonged Exposure + Placebo (PE/PLB)
Started (Treatment occurred weeks 0-24 and naturalistic follow-up continued through to week 52.) | 71 | 69 | 67
Completed | 50 | 49 | 40
Not Completed | 21 | 20 | 27
Not completed — Withdrawal by Subject | 4 | 5 | 10
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Lost to Follow-up | 16 | 15 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline + Enhanced Medication Management (SERT/EMM) | Prolonged Exposure + Sertraline (PE/SERT) | Prolonged Exposure + Placebo (PE/PLB) | Total
Number analyzed (Participants) | 71 | 69 | 67 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (8.2) | 35.1 (8.5) | 34.7 (8.3) | 34.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 8 | 27
  Male | 66 | 55 | 59 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 10 | 7 | 31
  Not Hispanic or Latino | 57 | 59 | 60 | 176
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 43 | 40 | 36 | 119
  Race: African American | 20 | 22 | 20 | 62
  Race: Other | 8 | 7 | 11 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71 | 69 | 67 | 207

OUTCOME MEASURES:

1. Primary Outcome: Posttraumatic Stress Disorder (PTSD) Symptoms as Measured by the Clinician Administered Posttraumatic Stress Disorder Scale (CAPS)
Description: Total Score; Range 0-136 with increasing PTSD severity as scores increase
Time Frame: 24 weeks
Population: All randomized patients who received treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sertraline + Enhanced Medication Management (SERT/EMM) | Prolonged Exposure + Sertraline (PE/SERT) | Prolonged Exposure + Placebo (PE/PLB)
Number analyzed (Participants) | 71 | 69 | 67
Scores on a scale | 41.7 (25.7) | 43.3 (27.2) | 51.5 (25.3)

2. Secondary Outcome: Patient Health Questionnaire-15
Description: PHQ-15; measures somatization and ranges from 0 to 30 and 0-9 is considered minimal/low, 10-14 is moderate, and 15-30 is severe
Time Frame: 24 weeks
Population: All Randomized patients who received treatment and had the measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sertraline + Enhanced Medication Management (SERT/EMM) | Prolonged Exposure + Sertraline (PE/SERT) | Prolonged Exposure + Placebo (PE/PLB)
Number analyzed (Participants) | 71 | 69 | 67
Scores on a scale | 8.6 (5.7) | 9.8 (5.7) | 10.5 (5.1)

ADVERSE EVENTS:
Time Frame: 52 weeks (24 Weeks of Treatment Phase and 28 weeks of follow-up)
Description: Individual descriptions were summarized to organ class
Arm/Group | Sertraline + Enhanced Medication Management (SERT/EMM) | Prolonged Exposure + Sertraline (PE/SERT) | Prolonged Exposure + Placebo (PE/PLB)
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/69 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/71 | 5/69 | 3/67
Other Adverse Events (participants affected / at risk) | 69/71 | 61/69 | 46/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline + Enhanced Medication Management (SERT/EMM) (N=71) | Prolonged Exposure + Sertraline (PE/SERT) (N=69) | Prolonged Exposure + Placebo (PE/PLB) (N=67)
Increased Suicidal Ideation (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2)
Increased Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Increased Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline + Enhanced Medication Management (SERT/EMM) (N=71) | Prolonged Exposure + Sertraline (PE/SERT) (N=69) | Prolonged Exposure + Placebo (PE/PLB) (N=67)
Cardiovascular (Cardiac disorders) | 2 (2) | 2 (2) | 4 (6)
Dermatological (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Endocrine (Endocrine disorders) | 6 (7) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 49 (94) | 34 (68) | 20 (39)
Genitourinary (Renal and urinary disorders) | 25 (36) | 17 (25) | 7 (7)
Hematological (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Muskuloskeletal (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9) | 3 (4)
Neurological (Nervous system disorders) | 27 (38) | 22 (29) | 14 (17)
Psychological (Psychiatric disorders) | 25 (40) | 24 (36) | 15 (25)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 10 (18) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No